CLINICAL TRIAL: NCT00470119
Title: Exercise Diet and Sex Hormones in Postmenopausal Women (NEW)
Brief Title: Effect of a Low-Calorie Diet and/or Exercise Program on Risk Factors for Developing Breast Cancer in Overweight or Obese Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Anne McTiernan, MD PhD, FHCRC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHS 1960.00; U54CA116847 (NIH); P50CA083636 (NIH); P30CA015704 (NIH); FHCRC-PHS-1960.00; FHCRC-1960; CDR0000544634 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer; Obesity; Weight Changes
Keywords: breast cancer; obesity; weight changes
MeSH Terms: conditions — Breast Neoplasms; Obesity; Body Weight Changes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention)
- Caloric Restriction (Other): Nutritionist-delivered weight loss intervention though diet modification with an aim of 10% weightloss over a year long intervention based on the DPP and LookAHEAD interventions. Participants meet with a nutritionist individually and in small groups. Participants receive general information about diet and behavior strategies such as self-monitoring, goal-setting, stimulus-control, problem-solving, and relapse-prevention training. Participants learn to set a calorie goal and a fat gram goal and how to achieve the goal calorie reduction. Meetings are held weekly during the first 6 months of the diet program but taper off over the course of the study.
  Interventions: Behavioral: behavioral dietary intervention
- Exercise Intervention (Other): Participants exercise 3 days per week under the supervision of a physiologist and 2 days per week independently at home, for a total of 5 exercise sessions (at least 45 minutes of moderate-intensity exercise per session) weekly over 12 months
  Interventions: Behavioral: Exercise intervention
- Caloric Restriction AND Exercise Intervention (Other): Combined caloric restriction & exercise intervention
  Interventions: Behavioral: behavioral dietary intervention; Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: behavioral dietary intervention — A group based modification of the DPP and LookAHEAD lifestyle programs with a goal of 10% weight loss
  Other Names: Weight Loss interventions
  Arms: Caloric Restriction; Caloric Restriction AND Exercise Intervention
Behavioral: Exercise intervention — Facility based and home-based exercise designed to increase moderate-to-vigorous aerobic activity in participants to 45 mins/day 5 days/week
  Arms: Caloric Restriction AND Exercise Intervention; Exercise Intervention

SUMMARY:
RATIONALE: A low-calorie diet and/or exercise program may help lower an overweight or obese postmenopausal woman's risk of developing breast cancer. It is not yet known whether a low-calorie diet and/or exercise program are more effective than no diet or exercise program in lowering an overweight or obese postmenopausal woman's risk of developing breast cancer.

PURPOSE: This randomized clinical trial is studying the effect of a low-calorie diet and/or exercise program on risk factors for developing breast cancer compared with no diet or exercise program in overweight or obese postmenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of a 1-year exercise intervention, reduced-calorie diet intervention, or a combined exercise and reduced-calorie diet intervention vs no intervention on serum estrone concentrations in overweight or obese postmenopausal women.

Secondary

* Compare the effects of these interventions on serum levels of estradiol and free estradiol in these participants.
* Compare the effects of these interventions on serum levels of testosterone and free testosterone in these participants.
* Compare the effects of these interventions on serum levels of sex hormone binding globulin in these participants.
* Compare the effects of these interventions on serum levels of insulin in these participants.
* Compare the effects of these interventions on serum levels of glucose in these participants.
* Compare the effects of these interventions on serum levels of c-peptide in these participants.
* Compare the effects of these interventions on serum levels of insulin-like growth factor I (IGF-1) in these participants.
* Compare the effects of these interventions on serum levels of insulin-like growth factor binding-protein-3 (IGFBP-3) in these participants.
* Compare the effects of these interventions on serum levels of c-reactive protein (CRP) in these participants.
* Compare the effects of these interventions on serum levels of serum amyloid protein A (SAA) in these participants.
* Compare the effects of these interventions on serum levels of interleukin-6 (IL-6) in these participants.
* Compare the effects of these interventions on serum levels of adiponectin in these participants.
* Compare the effects of these interventions on serum levels of leptin in these participants.
* Compare the effects of these interventions on serum levels of ghrelin in these participants.
* Compare the effects of these interventions on serum levels of Vitamin D in these participants.
* Compare the effects of these interventions on mammographic density in these participants.
* Compare the effects of these interventions on anthropometrics and body composition (i.e., weight, body mass index, total and percentage body fat, and waist and hip circumferences) in these participants.
* Compare the effects of these interventions on quality of life in these participants.
* Compare the effects of these interventions on numbers of leukocytes and neutrophiles in these participants.
* Compare the effects of these interventions on VO2max in these participants.

OUTLINE: This is a randomized study. Participants are stratified according to body mass index (< 30 vs ≥ 30). Participants are randomized to 1 of 4 intervention arms.

* Arm I (exercise program): Participants exercise 3 days per week under the supervision of a physiologist and 2 days per week independently at home, for a total of 5 exercise sessions (at least 45 minutes of moderate-intensity exercise per session) weekly over 12 months.
* Arm II (reduced-calorie diet): Participants meet with a nutritionist individually and in small groups. Participants receive general information about diet and behavior strategies such as self-monitoring, goal-setting, stimulus-control, problem-solving, and relapse-prevention training. Participants learn to set a calorie goal and a fat gram goal and how to achieve the goal calorie reduction. Meetings are held weekly during the first 6 months of the diet program but taper off over the course of the study.
* Arm III (exercise program and reduced-calorie diet): Participants meet with a physiologist and a nutritionist, as in arms I and II, and exercise and diet accordingly.
* Arm IV (control: delayed diet and exercise): Participants receive study materials on healthy diet and exercise at the end of the 12-month study period. In addition, participants are offered 2 months of group exercise training with a study physiologist and 4 group meetings with a nutritionist to learn about weight loss techniques and behavioral principles for achieving weight loss.

All participants undergo testing at baseline and periodically during study. Participants undergo blood collection for evaluation of serum levels of sex and metabolic hormones (e.g., estrone, estradiol, testosterone, free testosterone, and sex hormone binding globulin, radioimmunoassay and other immunoassays. Participants also undergo anthropometrics and body composition measurements and mammographic density assessment.

Participants complete questionnaires at baseline and at 6 and 12 months for assessment of diet and exercise. Quality of life (QOL) is measured at baseline and at 6 and 12 months using the Medical Outcomes Study 36-Item Short Form and the Impact of Weight on QOL questionnaire. Information on health habits, medical history, family history of breast cancer, and reproductive and menstrual history is also collected.

FINAL ACCRUAL: A total of 439 participants (118 in the caloric restriction arm, and 117 in both the CR+Exercise, and exercise only arm; and 87 in control arm) were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk for developing breast cancer due to any of the following lifestyle risk factors:

  * Lack of physical activity
  * Excess weight
  * Obesity
  * Weight gain over lifetime
* Body mass index > 25.0
* Physically able to undertake a moderate exercise or calorie reduction program
* No history of invasive or in situ breast cancer

PATIENT CHARACTERISTICS:

* Postmenopausal, defined by the absence of periods for the past 12 months
* Able to attend study clinic visits and classes, and undergo study measurements
* Able to fill out questionnaires and logs in English
* No moderate to high alcohol intake (more than 2 drinks per day)
* No concurrent smoking
* No invasive cancer within the past 10 years except simple basal cell or squamous cell carcinoma
* No diabetes mellitus

  * Fasting blood sugar < 126 mg/dL (on 2 occasions)
* Hematocrit 32-48%
* WBC 3,000-15,000/mm³
* Potassium 3.5-5.0 mEq/L
* Creatinine ≤ 2.0 mg/dL
* No abnormalities on screening physical that contraindicate study participation
* No contraindications for treadmill testing or entry into a training program, including any of the following:

  * Myocardial infarction within the past 6 months
  * Pulmonary edema
  * Myocarditis
  * Pericarditis
  * Unstable angina
  * Pulmonary embolism or deep vein thrombosis
  * Uncontrolled hypertension (i.e., blood pressure > 200/100 mm Hg)
  * Orthostatic hypotension
  * Moderate-to-severe aortic stenosis
  * Uncontrolled arrhythmia
  * Uncontrolled congestive heart failure
  * Third-degree heart block
  * Left bundle branch block
  * Thrombophlebitis
  * ST depression > 3 mm at rest
  * History of cardiac arrest or stroke
* Normal exercise treadmill testing (ETT)

  * Negative thallium or echo ETT required for patients with abnormal ETT (defined as ≥ 1.5 mm ST depression in > 1 lead within 1-minute recovery OR ≥ 1.1 mm ST depression in > 1 lead after 1-minute recovery OR reading of positive test by study doctor)
* No drug abuse
* No significant mental illness

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior and no concurrent menopausal hormone replacement therapy of any type, including vaginal route
* No concurrent participation in any other organized weight loss or exercise program
* No concurrent appetite suppressant medication
* No concurrent medications (e.g., weight-loss medications) likely to interfere with adherence to interventions or study outcomes

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2004-12; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Serum estrone concentrations as measured by radioimmunoassay | At baseline and 12 months timepoint

SECONDARY OUTCOMES:
Serum estradiol and free estradiol concentration as measured by radioimmunoassay | At baseline and 12 months timepoint
Testosterone and free testosterone as measured radioimmunoassay | At baseline and 12 months timepoint
Serum concentrations of Sex hormone binding globulin measured using immunoassays | At baseline and 12 months timepoint
Mammographic density measurements (i.e., percentage density and dense area of breast tissue) | At baseline and 12 months timepoint
Change in weight and body mass index (Anthropometrics) | At baseline and 12 months timepoint
Total and percentage body fat and body fat distribution (i.e., waist and hip circumferences) as measured by dual x-ray absorptiometry | At baseline and 12 months timepoint
Quality of life (assessed via questionnaires) | At baseline and 12 months timepoint
Change in daily caloric intake as measured by Food Frequency Questionnaire | At baseline and 12 months timepoint
Leukocyte and Neutrophil Counts | Baseline and 12 month timepoints
Serum concentrations of Insulin as measured radioimmunoassay | Baseline and 12 months
Serum concentrations of Glucose as measured radioimmunoassay | Baseline and 12 month timepoints
Serum concentrations of Insulin-like growth factor-1 | Baseline and 12 month timepoints
Serum concentrations of Insulin-like growth-factor binding protein-3 | Baseline and 12-month timepoints
Serum Vitamin D concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum ghrelin concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum C-reactive Protein (CRP) concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum concentrations of Serum Amyloid A (SAA) as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum interleukin-6 (IL-6) concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum adiponectin concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum leptin concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum androtenedione concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints
Serum c-peptide concentrations as measured by radioimmunoassay | Baseline and 12 month timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Anne McTiernan, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Duggan C, Tapsoba JD, Shivappa N, Harris HR, Hebert JR, Wang CY, McTiernan A. Changes in Dietary Inflammatory Index Patterns with Weight Loss in Women: A Randomized Controlled Trial. Cancer Prev Res (Phila). 2021 Jan;14(1):85-94. doi: 10.1158/1940-6207.CAPR-20-0181. Epub 2020 Aug 28. PMID 32859616
- [Derived] Mason C, de Dieu Tapsoba J, Duggan C, Wang CY, Alfano CM, McTiernan A. Eating behaviors and weight loss outcomes in a 12-month randomized trial of diet and/or exercise intervention in postmenopausal women. Int J Behav Nutr Phys Act. 2019 Nov 27;16(1):113. doi: 10.1186/s12966-019-0887-1. PMID 31775800
- [Derived] Duggan C, Tapsoba Jde D, Wang CY, McTiernan A. Dietary Weight Loss and Exercise Effects on Serum Biomarkers of Angiogenesis in Overweight Postmenopausal Women: A Randomized Controlled Trial. Cancer Res. 2016 Jul 15;76(14):4226-35. doi: 10.1158/0008-5472.CAN-16-0399. PMID 27417562
- [Derived] Habermann N, Makar KW, Abbenhardt C, Xiao L, Wang CY, Utsugi HK, Alfano CM, Campbell KL, Duggan C, Foster-Schubert KE, Mason CE, Imayama I, Blackburn GL, Potter JD, McTiernan A, Ulrich CM. No effect of caloric restriction or exercise on radiation repair capacity. Med Sci Sports Exerc. 2015 May;47(5):896-904. doi: 10.1249/MSS.0000000000000480. PMID 25160845
- [Derived] Duggan C, Xiao L, Terry MB, McTiernan A. No effect of weight loss on LINE-1 methylation levels in peripheral blood leukocytes from postmenopausal overweight women. Obesity (Silver Spring). 2014 Sep;22(9):2091-6. doi: 10.1002/oby.20806. Epub 2014 Jun 13. PMID 24930817
- [Derived] Imayama I, Alfano CM, Mason C, Wang C, Duggan C, Campbell KL, Kong A, Foster-Schubert KE, Blackburn GL, Wang CY, McTiernan A. Weight and metabolic effects of dietary weight loss and exercise interventions in postmenopausal antidepressant medication users and non-users: a randomized controlled trial. Prev Med. 2013 Nov;57(5):525-32. doi: 10.1016/j.ypmed.2013.07.006. Epub 2013 Jul 13. PMID 23859929
- [Derived] Mason C, Xiao L, Imayama I, Duggan CR, Foster-Schubert KE, Kong A, Campbell KL, Wang CY, Villasenor A, Neuhouser ML, Alfano CM, Blackburn GL, McTiernan A. Influence of diet, exercise, and serum vitamin d on sarcopenia in postmenopausal women. Med Sci Sports Exerc. 2013 Apr;45(4):607-14. doi: 10.1249/MSS.0b013e31827aa3fa. PMID 23190588
- [Derived] Mason C, Foster-Schubert KE, Imayama I, Xiao L, Kong A, Campbell KL, Duggan CR, Wang CY, Alfano CM, Ulrich CM, Blackburn GL, McTiernan A. History of weight cycling does not impede future weight loss or metabolic improvements in postmenopausal women. Metabolism. 2013 Jan;62(1):127-36. doi: 10.1016/j.metabol.2012.06.012. Epub 2012 Aug 14. PMID 22898251
- [Derived] Mason C, Foster-Schubert KE, Imayama I, Kong A, Xiao L, Bain C, Campbell KL, Wang CY, Duggan CR, Ulrich CM, Alfano CM, Blackburn GL, McTiernan A. Dietary weight loss and exercise effects on insulin resistance in postmenopausal women. Am J Prev Med. 2011 Oct;41(4):366-75. doi: 10.1016/j.amepre.2011.06.042. PMID 21961463
- [Derived] Mason C, Xiao L, Imayama I, Duggan CR, Bain C, Foster-Schubert KE, Kong A, Campbell KL, Wang CY, Neuhouser ML, Li L, W Jeffery R, Robien K, Alfano CM, Blackburn GL, McTiernan A. Effects of weight loss on serum vitamin D in postmenopausal women. Am J Clin Nutr. 2011 Jul;94(1):95-103. doi: 10.3945/ajcn.111.015552. Epub 2011 May 25. PMID 21613554